CLINICAL TRIAL: NCT03341130
Title: Determinants of Occlusal Changes in Oral Appliance Treatment of OSA - A Randomized Controlled Trial
Brief Title: Determinants of Tooth Movement in Oral Appliance Treatment of OSA.
Acronym: TACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Université de Montréal (Other); Laval University (Other)
Responsible Party: Principal Investigator, Benjamin Pliska, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F17-00320
Record Dates: First submitted 2017-11-02; First posted 2017-11-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Mandibular Advancement Splint; Oral Appliance; Treatment; Repositioning Splint
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analysis of primary outcomes will be performed by an examiner blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Treatment Group (Experimental): The treatment group will will be treated a mandibular advancement oral appliance following standard practices. The treatment group will also receive a mandibular repositioning splint to wear in the mornings for a minimum of 1 hour following removal of their mandibular advancement oral appliance, in an effort to reduce the side effects resulting from use of the mandibular advancement oral appliance.
  Interventions: Device: Mandibular Repositioning Splint; Device: Mandibular Advancement Oral Appliance
- Positive Control Group (Experimental): The positive control group will will be treated a mandibular advancement oral appliance following standard practices. The positive control group will not receive any additional oral appliances. Side effects resulting from use of the mandibular advancement oral appliance will be managed using standard practices, including jaw stretching exercises as needed for comfort.
  Interventions: Device: Mandibular Advancement Oral Appliance
- Negative Control Group (No Intervention): The negative control group is comprised of 15 healthy individuals recruited specifically from faculty members at the UBC Faculty of Dentistry. This group will undergo the same clinical data collection as the treatment group and the negative control group but will not receive any treatment.

INTERVENTIONS:
Device: Mandibular Repositioning Splint — The Morning Repositioner is a hands-free bite deprogrammer designed to help return the patient's jaw back to its pre-treatment centric position.
  Other Names: Morning Repositioner; Morning Aligner
  Arms: Treatment Group
Device: Mandibular Advancement Oral Appliance — Mandibular Advancement Oral Appliances are dental splints used to keep the jaw in an advanced position, opening the upper airway during sleep.
  Other Names: OAM; MAS
  Arms: Positive Control Group; Treatment Group

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep related breathing disorder, affecting approximately 10% of adults. Mandibular advancement oral appliances (OAM) are an effective treatment for OSA, however, long term use has shown to lead to changes in teeth positioning and jaw alignment (bite changes), which has resulted in some patients stopping treatment.

It is becoming common clinical practice for doctors to prescribe the use of repositioning splints to help reduce the bite changes associated with using OAM. However, this has not been studied in a clinical trial.

This study will compare the bite changes between patients using OAM alone against patients using a morning repositioning splint in addition to OAM. Other variables, such as oral health, the size of mandibular advancement, and treatment adherence will also be measured to determine if they have an effect on the bite changes associated with OAM use.

By understanding the key the factors that influence the bite changes associated with OAM use and potentially validating a technique to reduce these changes, this study will improve the clinical practice of Dental Sleep Medicine, leading to improved health outcomes for OSA patients.

DETAILED DESCRIPTION:
Mandibular advancement oral appliances (OAM) are an effective treatment for obstructive sleep apnea (OSA). However, prolonged OAM treatment leads to significant changes in occlusion for the majority of patients. As such it is not uncommon to find changes in occlusion and the resulting decrease in quality of life in long-term users of oral appliances to be cited as a reason for discontinuing OAM treatment. Understanding the determinants of occlusal changes and clinical strategies to minimize or prevent them are essential to the practice of Dental Sleep Medicine, where treatment success is predicated on high levels of adherence.

Morning Repositioners or alternative oral appliances/splints that counteract the muscle splinting of the mandible in a forward postured position have been advocated by some practitioners as a means of minimizing the occlusal changes associated with OAM treatment. However, this has not been studied in a prospective clinical trial.

The proposed study is a single-blinded prospective randomized controlled trial at three clinical centers, with the specific aim of assessing the effectiveness of mandibular repositioning splint use on minimizing the occlusal changes associated with OAM treatment. Secondary aims include also determining the effects of periodontal disease, treatment adherence, and magnitude of mandibular advancement on occlusal changes associated with OAM treatment.

90 OSA patients will receive OAM treatment following standard practices. A titration period of two months will be used to adjust the position of mandibular advancement for each patient, which will involve clinical follow-up visits at a minimum of 1 week, 1 month and 2 months after initiation of OAM treatment. Each participant will be randomly assigned to either the treatment or control group. The treatment group will receive a mandibular repositioning splint to wear for a minimum of 1 hour in the mornings following removal of OAM. A positive control group will receive no additional splint, and but will be managed using standard practices, including jaw stretching exercises as needed. A second negative control group consisting of 15 healthy adults not undergoing any oral appliance treatment will also be included.

Prior to receiving treatment, participants will undergo a baseline assessment where demographic, anthropometric, and specific periodontal health data will be collected. All measurements will be repeated at a minimum of 18 and 36 months after appliance insertion, with routine follow-up appointments and adherence data collected every six months.

To directly address the primary aim of this study, occlusal variables will be measured by a combination of methods including analysis of digitized dental models, cephalometric analysis and intra-oral radiography bone level measurements. Secondary outcome variables to assess the effectiveness of morning mandibular repositioning splint therapy will include average OAM adherence (hours/night), quality of life (Functional Outcomes of Sleep Questionnaire, FOSQ), and change in mandibular incisor root length and attachment loss. Adherence will be measured by compliance monitors embedded in the oral appliance and mandibular repositioning splints.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive (have never used an oral appliance as treatment for OSA);
* Age 25 - 65 years old, who are able to freely provide informed consent;
* Body Mass Index (BMI) ≤ 35;
* 8 or more teeth per arch to support treatment with OAM;
* Apnea-Hypopnea Index (AHI) within the range 5≤AHI≤50 documented with polysomnography in the last 2 years ***OR***
* Respiratory Disturbance Index (RDI) within the range 20 ≤ RDI ≤ 50 documented with level III portable sleep test ***OR***
* Oxygen Desaturation Index (ODI) ≥ 10

Exclusion Criteria:

* Extensive periodontal disease with significant tooth mobility;
* Inability to protrude jaw;
* Insufficient vertical opening to accommodate treatment with OAM;
* Pregnancy (if a participant becomes pregnant during the trial, the participant will be withdrawn from the study).
* Uncontrolled congestive heart failure (defined as a prior clinical diagnosis, an ejection cut-off of 40% or clinical sign in the opinion of a primary care physician or cardiologist) that makes it unsafe in the opinion of the investigators for the subject to participate in the trial;
* Coronary artery disease unless stable for at least 6 months and considered by the investigators to have a stable disease;
* Any history of angina, myocardial infarction or stroke;
* Any history of major depressive disorder along with current moderate-severe disease;
* Active cancer management (unless in remission for more than 1 year);
* Known renal failure (with need for dialysis)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Overjet | Data collected at 0, 18 and 36 months after appliance insertion.
  The change in the extent of horizontal (anterior-posterior) overlap of the maxillary central incisors over the mandibular central incisors, measured from digital dental model analysis.

SECONDARY OUTCOMES:
Treatment Adherence | Data collected every 6 months after treatment commencement, up to 36 months.
  Adherence will be measured by the DentiTrac smart chip (Braebon Medical Corporation, Kanata, Canada) embedded in the oral appliance and mandibular repositioning splints. The adherence will be measured in hours per night and nights per week.
Quality of Life using Functional Outcomes of Sleep Questionnaire (FOSQ-10) | Data collected at 0, 1, 2, 18 and 36 months after appliance insertion.
  FOSQ-10 measures functional status and difficulty in performing everyday activities via 10 questions. The range of scores for any question is from 1 to 4. There is also a 0 score option for participants who do not engage in a particular activity for other reasons, in which case the question will be excluded. There are 5 subscales that measure: general productivity, activity level, vigilance, social outcomes, and intimacy and sexual relationships. To obtain the total score, a mean-weighted item score is computed for those subscales with more than one item. To calculate a mean-weighted item score calculate the mean of the answered items with responses > 1 for each subscale. The total score is then derived by calculating the mean of the subscale scores and multiplying that mean by five. Total score ranges between 5 and 20. Higher scores indicate better functional status.
Daytime Sleepiness | Data collected at 0, 1, 2, 18 and 36 months after appliance insertion.
  Evaluation of OSA specific fatigue using Epworth Sleepiness Scale (ESS) questionnaire. ESS measures daytime sleepiness via 8 questions that ask about daytime sleepiness during common everyday conditions. The potential range of scores for any questions is from 0 to 3. Higher values represent worse outcomes. Their are no subscales for ESS. The answers to the questions are all summed up. Total score ranges between 0 and 24. A score above 10 indicates daytime sleepiness with higher scores indicating more sleepiness.
Change in Overbite | Data collected at 0, 18 and 36 months after appliance insertion.
  Using digital dental model analysis to evaluate the change in the extent of vertical (superior-inferior) overlap of the maxillary central incisors over the mandibular central incisors, measured relative to the incisal edges.
Dental Crowding | Data collected at 0, 18 and 36 months after appliance insertion.
  Changes in dental crowding, measured by digital dental model analysis.
Intermolar Distance | Data collected at 0, 18 and 36 months after appliance insertion.
  Changes in distance between molars, measured by digital dental model analysis.
Intercanine Distance | Data collected at 0, 18 and 36 months after appliance insertion.
  Changes in distance between canines, measured by digital dental model analysis.
Posterior Occlusal Changes | Data collected at 0, 18 and 36 months after appliance insertion.
  Changes in the number of posterior teeth with open occlusal contacts, measured from digital dental model analysis.
Anterior Occlusal Changes | Data collected at 0, 18 and 36 months after appliance insertion.
  Change in the number of anterior teeth in crossbite, measured from digital dental model analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Pliska, DDS, Principal Investigator — University British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada